CLINICAL TRIAL: NCT02153411
Title: Evaluation of aSthma Management in Middle EAst Adult Population
Brief Title: Multicentric, Transversal, Descriptive, Epidemiological Study on the Management of Asthma in Asthmatic Middle East Adult Population
Acronym: ESMAA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-RME-XXX-2014/1; NIS-RME-XXX-2014/1 (Registry Identifier: NIS Registry)
Record Dates: First submitted 2014-05-30; First posted 2014-06-03 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
Keywords: Asthma control
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 8645 asthmatic patients: Men and women, 18 years of age and older. Asthmatic since at least one year before inclusion. Patient's informed consent obtained.

SUMMARY:
Descriptive study on the management of asthma in asthmatic Middle East adult population : Algeria,Egypt, Irak,Iran, Jordan, Koweit, Lebanon, Qatar,Saudi,Tunisia, UAE

DETAILED DESCRIPTION:
Multicentric, transversal, descriptive, epidemiological study, conducted in a random sample of general practitioner and medical specialist (Pulmonologist and/or allergologist) in the public and the private sector.

ELIGIBILITY:
Inclusion Criteria:

Men and women, 18 years of age and older. Asthmatic since at least one year before inclusion. Patient's informed consent obtained.

Exclusion Criteria:

* Patient concurrently participating to another study. Patient with concomitant pulmonary disease. Patient with psychiatric disorders. Patient consulting for an asthma attack

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthmatic since at least one year before inclusion. Patient's informed consent obtained.
Sampling Method: Non-Probability Sample
Enrollment: 7294 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Asthma control | Up to 1 year
  Daytime symptoms Limitation of activities Nocturnal symptoms / awakening Need for reliever /rescue treatment Lung function (PEF or FEV)

SECONDARY OUTCOMES:
general and sociodemographic patient's characteristics | up to 1 year
  sex, age, BMI, educational level, occupation, comorbidities, smoking status, and social security coverage.
Identify predictive factors of asthma control, | UP to 1 year
  such as age, sex, BMI, smoking status, adherence to treatment, asthma history, comorbidity.
asthma control level | Up to 4 weeks
  Asthma control test questionnaire : activities at work,breathless,asthma symptoms (wheezing, coughing, chest tightness, shortness of breath;use of rescue inhaler or taken a nebulizer treatment ,asthma assessment

CONTACTS AND LOCATIONS:
Locations (98):
- Algeria (37):
  - Research Site, Ain Naadja, Nis-rme-xxx-2014/1
  - Research Site, Aïn Beïda, Nis-rme-xxx-2014/1
  - Research Site, Algiers, Nis-rme-xxx-2014/1
  - Research Site, Annaba, Nis-rme-xxx-2014/1
  - Research Site, Azzaba, Nis-rme-xxx-2014/1
  - Research Site, Bab Ezzouar, Nis-rme-xxx-2014/1
  - Research Site, Babez, Nis-rme-xxx-2014/1
  - Research Site, Batna City, Nis-rme-xxx-2014/1
  - Research Site, Bāb al-Wādī, Nis-rme-xxx-2014/1
  - Research Site, Béjaïa, Nis-rme-xxx-2014/1
  - Research Site, Birkhadem, Nis-rme-xxx-2014/1
  - Research Site, Blida, Nis-rme-xxx-2014/1
  - Research Site, Bordj Bou Arreridj, Nis-rme-xxx-2014/1
  - Research Site, Bordj Menail, Nis-rme-xxx-2014/1
  - Research Site, Bouïra, Nis-rme-xxx-2014/1
  - Research Site, Bouzarea, Nis-rme-xxx-2014/1
  - Research Site, Constantine, Nis-rme-xxx-2014/1
  - Research Site, El Eulma, Nis-rme-xxx-2014/1
  - Research Site, Essania, Nis-rme-xxx-2014/1
  - Research Site, Gouraya, Nis-rme-xxx-2014/1
  - Research Site, Lakhdaria, Nis-rme-xxx-2014/1
  - Research Site, Larbaâ, Nis-rme-xxx-2014/1
  - Research Site, M'Sila, Nis-rme-xxx-2014/1
  - Research Site, Mascara, Nis-rme-xxx-2014/1
  - Research Site, Meftah, Nis-rme-xxx-2014/1
  - Research Site, Mila, Nis-rme-xxx-2014/1
  - Research Site, Misserghin, Nis-rme-xxx-2014/1
  - Research Site, Mostaghanem, Nis-rme-xxx-2014/1
  - Research Site, Oran, Nis-rme-xxx-2014/1
  - Research Site, Ouled Beni Messous, Nis-rme-xxx-2014/1
  - Research Site, Rouiba, Nis-rme-xxx-2014/1
  - Research Site, Sétif, Nis-rme-xxx-2014/1
  - Research Site, Sidi Bel Abbes, Nis-rme-xxx-2014/1
  - Research Site, Tiaret, Nis-rme-xxx-2014/1
  - Research Site, Tipasa, Nis-rme-xxx-2014/1
  - Research Site, Tizi Ouzou, Nis-rme-xxx-2014/1
  - Research Site, Zeralda, Nis-rme-xxx-2014/1
- Egypt (11):
  - Research Site, Alexandria, Nis-rme-xxx-2014/1
  - Research Site, Cairo, Nis-rme-xxx-2014/1
  - Research Site, Domyat - Delta, Nis-rme-xxx-2014/1
  - Research Site, Giza - Cairo, Nis-rme-xxx-2014/1
  - Research Site, Ismalia - Delta, Nis-rme-xxx-2014/1
  - Research Site, Mansoura - Delta, Nis-rme-xxx-2014/1
  - Research Site, Menofia - Delta, Nis-rme-xxx-2014/1
  - Research Site, Menoufia - Delta, Nis-rme-xxx-2014/1
  - Research Site, Portsaid - Delta, Nis-rme-xxx-2014/1
  - Research Site, Tanta - Delta, Nis-rme-xxx-2014/1
  - Research Site, Zagazig - Delta, Nis-rme-xxx-2014/1
- Iran (11):
  - Research Site, Ahvāz, Nis-rme-xxx-2014/1
  - Research Site, Isfahan, Nis-rme-xxx-2014/1
  - Research Site, Karaj, Nis-rme-xxx-2014/1
  - Research Site, Kerman, Nis-rme-xxx-2014/1
  - Research Site, Mashhad, Nis-rme-xxx-2014/1
  - Research Site, Rasht, Nis-rme-xxx-2014/1
  - Research Site, Sari, Nis-rme-xxx-2014/1
  - Research Site, Shiraz, Nis-rme-xxx-2014/1
  - Research Site, Tabriz, Nis-rme-xxx-2014/1
  - Research Site, Tehran, Nis-rme-xxx-2014/1
  - Research Site, Yazd, Nis-rme-xxx-2014/1
- Iraq (7):
  - Research Site, Baghdad, Nis-rme-xxx-2014/1
  - Research Site, Basra, Nis-rme-xxx-2014/1
  - Research Site, Erbil, Nis-rme-xxx-2014/1
  - Research Site, Hillah, Nis-rme-xxx-2014/1
  - Research Site, Manşūrīyah, Nis-rme-xxx-2014/1
  - Research Site, Najaf, Nis-rme-xxx-2014/1
  - Research Site, Sulaimania, Nis-rme-xxx-2014/1
- Jordan (6):
  - Research Site, Amman, Nis-rme-xxx-2014/1
  - Research Site, Irbid, Nis-rme-xxx-2014/1
  - Research Site, Madaba, Nis-rme-xxx-2014/1
  - Research Site, Russeifa, Nis-rme-xxx-2014/1
  - Research Site, Salt, Nis-rme-xxx-2014/1
  - Research Site, Zarqa, Nis-rme-xxx-2014/1
- Kuwait (3):
  - Research Site, Kuwait City, Nis-rme-xxx-2014/1
  - Research Site, Kuwait City, Nis-rme-xxx-2014/2
  - Research Site, Kuwait City, Nis-rme-xxx-2014/5
- Lebanon (10):
  - Research Site, Bkaa, Nis-rme-xxx-2014/1
  - Research Site, Chweifat, Nis-rme-xxx-2014/1
  - Research Site, Dahieh, Nis-rme-xxx-2014/1
  - Research Site, East Beirut, Nis-rme-xxx-2014/1
  - Research Site, Keserwen, Nis-rme-xxx-2014/1
  - Research Site, Maten, Nis-rme-xxx-2014/1
  - Research Site, North Beirut, Nis-rme-xxx-2014/1
  - Research Site, South Beirut, Nis-rme-xxx-2014/1
  - Research Site, South Metn, Nis-rme-xxx-2014/1
  - Research Site, West Beirut, Nis-rme-xxx-2014/1
- Research Site, Doha, Nis-rme-xxx-2014/1, Qatar
- Saudi Arabia (5):
  - Research Site, Al Hadā, Nis-rme-xxx-2014/1
  - Research Site, Dammam, Nis-rme-xxx-2014/1
  - Research Site, Jeddah, Nis-rme-xxx-2014/1
  - Research Site, Khobar, Nis-rme-xxx-2014/1
  - Research Site, Riyadh, Nis-rme-xxx-2014/1
- Tunisia (3):
  - Research Site, Sfax, Nis-rme-xxx-2014/1
  - Research Site, Sousse, Nis-rme-xxx-2014/1
  - Research Site, Tunis, Nis-rme-xxx-2014/1
- United Arab Emirates (4):
  - Research Site, Abu Dhabi, Nis-rme-xxx-2014/1
  - Research Site, Al Ain City, Nis-rme-xxx-2014/1
  - Research Site, Dubai, Nis-rme-xxx-2014/1
  - Research Site, Sharjah city, Nis-rme-xxx-2014/1

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3007&filename=CSRsynopsis.pdf